CLINICAL TRIAL: NCT07406555
Title: Differences in C-Reactive Protein Levels Between Traumatic Brain Injury Patients Receiving Dexmedetomidine and Those Not Receiving Dexmedetomidine Undergoing Craniotomy at Prof. Dr. Margono Soekarjo Regional General Hospital, Purwokerto
Brief Title: Comparison of C-Reactive Protein Levels in Traumatic Brain Injury Patients Undergoing Craniotomy With and Without Dexmedetomidine
Acronym: DEX-CRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Jenderal Soedirman (Other)
Responsible Party: Principal Investigator, Adrian Nugraha Putra, Principal Investigator, Universitas Jenderal Soedirman
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 146/KEPK/PE/XII/2025
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Brain Injury
Keywords: Dexmedetomidine; C-Reactive Protein; Craniotomy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Intervention Model Description: A parallel-group interventional study comparing C-Reactive Protein (CRP) levels between patients receiving intravenous Dexmedetomidine and a control group (standard care) during craniotomy for traumatic brain injury
Who Masked: Participant, Care Provider, Investigator
Masking Description: A parallel-group interventional study to compare the effect of Dexmedetomidine administration on C-Reactive Protein (CRP) levels in traumatic brain injury patients undergoing craniotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): Patients undergoing craniotomy for traumatic brain injury who receive Dexmedetomidine administration.
  Interventions: Drug: Dexmedetomidine
- control (Active Comparator): Patients undergoing craniotomy for traumatic brain injury receiving Sufentanyl as the standard analgesic/sedative agent.
  Interventions: Drug: Sufentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous administration of Dexmedetomidine to evaluate its effect on inflammatory markers (CRP)
  Arms: Dexmedetomidine Group
Drug: Sufentanyl — Intravenous administration of Sufentanyl as an active comparator in the control group
  Arms: control

SUMMARY:
Traumatic brain injury is a major cause of morbidity and mortality and is often associated with a systemic inflammatory response after surgery. C-reactive protein (CRP) is a commonly used biomarker to assess inflammation. Dexmedetomidine is an anesthetic adjuvant that may have anti-inflammatory effects.

This study aims to compare C-reactive protein levels in traumatic brain injury patients undergoing craniotomy who receive dexmedetomidine with those who do not receive dexmedetomidine. The study is conducted at Prof. Dr. Margono Soekarjo Regional General Hospital, Purwokerto. The results of this study are expected to provide information on the potential effect of dexmedetomidine on postoperative inflammatory response in traumatic brain injury patients.

DETAILED DESCRIPTION:
This study is an interventional study conducted in traumatic brain injury patients undergoing craniotomy at Prof. Dr. Margono Soekarjo Regional General Hospital, Purwokerto. Eligible patients are divided into two groups: patients who receive dexmedetomidine as part of perioperative management and patients who do not receive dexmedetomidine.

C-reactive protein levels are measured as an indicator of systemic inflammatory response. The primary objective of the study is to compare CRP levels between the two groups. Data are collected from medical records and laboratory examinations and analyzed to evaluate differences in inflammatory response between patients receiving dexmedetomidine and those not receiving dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years to ≤ 60 years
* Patients with secondary brain injury with onset ≥ 6 hours
* Patients with a GCS score > 6 undergoing emergency and elective craniotomy
* American Society of Anesthesiologists (ASA) physical status ≥ II
* Body mass index > 17 kg/m² and < 30 kg/m²

Exclusion Criteria:

* Patients with head injury onset < 6 hours
* Patients with signs of systemic shock
* Patients or family members who refuse to participate
* Patients with a history of allergy to dexmedetomidine, sevoflurane, and/or sufentanil
* Patients with a history of active infection or sepsis
* Patients who have received massive blood transfusion prior to surgery
* Patients with autoimmune diseases
* Patients with active malignancy
* Patients with a history of chemotherapy
* Patients with a history of hepatic dysfunction, indicated by elevated alanine aminotransferase (ALT/SGPT) levels above the normal reference range (7-56 U/L)
* Patients with a history of long-term corticosteroid therapy
* Patients with a history of neuropsychiatric disorders and cognitive impairment
* Patients with a history of pre-existing cardiovascular disease
* Patients with a history of coagulation disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-10-27 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Change in C-Reactive Protein (CRP) Levels | Baseline (Pre-operative), 6 hours and 24 hours post-operative
  Serum CRP levels measured to assess the inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Nugraha Putra, Principal Investigator — Universitas Jenderal Soedirman
Locations (1):
- RSUD Prof. Dr. Margono Soekarjo, Purwokerto, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao, Y. et al. (2020) 'Mechanisms of Dexmedetomidine in Neuropathic Pain', Frontiers in Neuroscience. Frontiers Media S.A. Available at: https://doi.org/10.3389/fnins.2020.00330
- [Background] Xu, J. and Xiao, Q. (2022) 'Assessment of the effects of dexmedetomidine on outcomes of traumatic brain injury using propensity score analysis', BMC Anesthesiology, 22(1). Available at: https://doi.org/10.1186/s12871-022-01822-2.
- [Background] Wiles, M.D. (2022) 'Management of traumatic brain injury: a narrative review of current evidence', Anaesthesia. John Wiley and Sons Inc, pp. 102-112. Available at: https://doi.org/10.1111/anae.15608
- [Background] Weerink, M.A.S. et al. (2017) 'Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine', Clinical Pharmacokinetics, 56(8), pp. 893-913. Available at: https://doi.org/10.1007/s40262-017-0507-7
- [Background] Vitali, M. et al. (2023) 'Decompressive Craniectomy in Severe Traumatic Brain Injury: The Intensivist's Point of View', Diseases, 11(1). Available at: https://doi.org/10.3390/diseases11010022
- [Background] Thapa, K. et al. (2021) 'Traumatic Brain Injury: Mechanistic Insight on Pathophysiology and Potential Therapeutic Targets', Journal of Molecular Neuroscience, 71(9), pp. 1725-1742. Available at: https://doi.org/10.1007/s12031-021-01841-7
- [Background] Slupe, A.M. and Kirsch, J.R. (2018) 'Effects of anesthesia on cerebral blood flow, metabolism, and neuroprotection', Journal of Cerebral Blood Flow and Metabolism, 38(12), pp. 2192-2208. Available at: https://doi.org/10.1177/0271678X18789273
- [Background] Sakti, S., Kriswidyatomo, P. and Sumartono, C. (2025) 'The Effect of Dexmedetomidine on Post-Operative C-Reactive Protein Levels in Patients Undergoing Brain Tumor Resection: A Literature Review', Vascular and Endovascular Review, 8. Available at: www.VERjournal.com
- [Background] Randall, Z.D. et al. (2022) 'Demographic, behavioral, dietary, and clinical predictors of high-sensitivity C-reactive protein: The National Health and Nutrition Examination Surveys (NHANES)', American Heart Journal Plus: Cardiology Research and Practice, 21. Available at: https://doi.org/10.1016/j.ahjo.2022.100196
- [Background] Ng, S.Y. and Lee, A.Y.W. (2019) 'Traumatic Brain Injuries: Pathophysiology and Potential Therapeutic Targets', Frontiers in Cellular Neuroscience, 13. Available at: https://doi.org/10.3389/fncel.2019.00528
- [Background] Murdoch, I., Surda, P. and Nguyen-Lu, N. (2021) 'Anaesthesia for rhinological surgery', BJA Education, 21(6), pp. 225-231. Available at: https://doi.org/10.1016/j.bjae.2021.02.004
- [Background] Liu, X. et al. (2021) 'Recent Advances in the Clinical Value and Potential of Dexmedetomidine', Journal of Inflammation Research, 14, pp. 7507-7527. Available at: https://doi.org/10.2147/JIR.S346089
- [Background] Li, Y. et al. (2015) 'Effect of dexmedetomidine on early postoperative cognitive dysfunction and peri-operative inflammation in elderly patients undergoing laparoscopic cholecystectomy', Experimental and Therapeutic Medicine, 10(5), pp. 1635-1642. Available at: https://doi.org/10.3892/etm.2015.2726
- [Background] Kim, H. (2023) 'Anesthetic management of the traumatic brain injury patients undergoing non-neurosurgery', Anesthesia and Pain Medicine, 18(2), pp. 104-113. Available at: https://doi.org/10.17085/apm.23017
- [Background] Huang, Y. et al. (2022) 'Comparing the Effect of Dexmedetomidine and Midazolam in Patients with Brain Injury', Brain Sciences, 12(6). Available at: https://doi.org/10.3390/brainsci12060752
- [Background] Huang, C.Y. et al. (2024) 'Assessing the Predictive Utility of the C-Reactive Protein-to-Lymphocyte Ratio for Mortality in Isolated Traumatic Brain Injury: A Single-Center Retrospective Analysis', Diagnostics, 14(18). Available at: https://doi.org/10.3390/diagnostics14182065
- [Background] Hu, Y. et al. (2022) 'The neuroprotective effect of dexmedetomidine and its mechanism', Frontiers in Pharmacology, 13(September), pp. 1-15. Available at: https://doi.org/10.3389/fphar.2022.965661
- [Background] Hosseininejad, S.M. et al. (2023) 'C-Reactive Protein and D-Dimer as Prognostic Markers for Clinical Outcomes in Patients with Mild Traumatic Brain Injury: A Cross-Sectional Study', Journal compilation © 2023 Trauma Research Center, Shiraz University of Medical Sciences Hosseininejad SM et al. Bull Emerg Trauma, 11(3), pp. 119-124. Available at: https://doi.org/10.30476/BEAT.2023.98573.1435
- [Background] Hatfield, J. et al. (2024) 'Safety, Efficacy, and Clinical Outcomes of Dexmedetomidine for Sedation in Traumatic Brain Injury: A Scoping Review', Journal of Neurosurgical Anesthesiology, 36(2), pp. 101-108. Available at: https://doi.org/10.1097/ANA.0000000000000907
- [Background] Haarbauer-Krupa, J. et al. (2021) 'Epidemiology of Chronic Effects of Traumatic Brain Injury', Journal of Neurotrauma, 38(23), pp. 3235-3247. Available at: https://doi.org/10.1089/neu.2021.0062
- [Background] Feng, X. et al. (2021) 'Dexmedetomidine alleviates early brain injury following traumatic brain injury by inhibiting autophagy and neuroinflammation through the ROS/Nrf2 signaling pathway', Molecular Medicine Reports, 24(3). Available at: https://doi.org/10.3892/mmr.2021.12300
- [Background] Ding, M. et al. (2019) 'Dexmedetomidine reduces inflammation in traumatic brain injury by regulating the inflammatory responses of macrophages and splenocytes', Experimental and Therapeutic Medicine [Preprint]. Available at: https://doi.org/10.3892/etm.2019.7790
- [Background] Dewan, M.C. et al. (2019) 'Estimating the global incidence of traumatic brain injury', Journal of Neurosurgery, 130(4), pp. 1080-1097. Available at: https://doi.org/10.3171/2017.10.JNS17352
- [Background] Department of Nutrition for Health and Development World Health Organization. (2014) C-reactive protein concentrations as a marker of inflammation or infection for interpreting biomarkers of micronutrient status, Geneva. Available at: http://apps.who.int/iris/bitstream/10665/133708/1/WHO
- [Background] Dahlan, M.S. (2019) Besar Sampel dalam Penelitian Kedokteran dan Kesehatan. Jakarta: Epidemiologi Indonesia.
- [Background] Crowe, G., Atterton, B. and Moran, L. (2022) 'Perioperative Applications of Dexmedetomidine', Anaesthesia Tutorial of The Week [Preprint]. Available at: https://resources.wfsahq.org/anaesthesia-tutorial-of-the-week/.
- [Background] Chen, R. et al. (2021) 'The Anti-inflammatory Effect of Dexmedetomidine Administration on Patients Undergoing Intestinal Surgery: A Randomized Study', Drugs in R and D, 21(4), pp. 445-453. Available at: https://doi.org/10.1007/s40268-021-00368-x.
- [Background] Brodier, E.A. and Cibelli, M. (2021) 'Postoperative cognitive dysfunction in clinical practice', BJA Education. Elsevier Ltd, pp. 75-82. Available at: https://doi.org/10.1016/j.bjae.2020.10.004
- [Background] Bastian, B., Sari, I. and Pratama, F.P. (2022) 'Analysis of C-Reactive Protein (CRP) Levels in Venous and Capillary Blood Samples with Immunoturbidimetric Methods', Medicra (Journal of Medical Laboratory Science/Technology), 5(1), pp. 1-5. Available at: https://doi.org/10.21070/medicra.v5i1.1622.
- [Background] Bafna, U. et al. (2021) 'Comparison of hypotensive properties of dexmedetomidine versus clonidine for induced hypotension during functional endoscopic sinus surgery: A randomised, double-blind interventional study', Indian Journal of Anaesthesia, 65(8), pp. 579-585. Available at: https://doi.org/10.4103/ija.IJA_57_21.
- [Background] Ayala J, Smith A, F.D. (2006) 'C-reactive protein levels following cardiac surgery in adults', European Journal of Anaesthesiology | EJA, 23, p. 758.
- [Background] Ali, S. et al. (2023) 'Role of C-reactive protein in disease progression, diagnosis and management', Discoveries, 11(4), p. e179. Available at: https://doi.org/10.15190/d.2023.18.
- [Background] Akashi, N. et al. (2021) 'Cardiovascular and renal effects of constant rate infusions of remifentanil, dexmedetomidine and their combination in dogs anesthetized with sevoflurane', Journal of Veterinary Medical Science, 83(2), pp. 285-296. Available at: https://doi.org/10.1292/jvms.20-0457.